CLINICAL TRIAL: NCT03059823
Title: A Phase 1 Study of the Safety, Tolerability, and Pharmacokinetics of INCMGA00012 in Patients With Advanced Solid Tumors
Brief Title: A Phase 1 Study of INCMGA00012 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCMGA 0012-101; 2017-000865-63 (EudraCT Number)
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced Solid Tumors; Metastatic Solid Tumors
Keywords: Solid tumors; Metastatic cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation-Q2W (Experimental): INCMGA00012 treatment once every 2 weeks.
  Interventions: Drug: retifanlimab
- Dose Escalation- Q3W (Experimental): INCMGA00012 treatment once every 3 weeks.
  Interventions: Drug: retifanlimab
- Dose Escalation- Q4W (Experimental): INCMGA00012 treatment once every 4 weeks.
  Interventions: Drug: retifanlimab
- Expansion Cohort (Experimental): INCMGA00012 treatment for locally advanced or metastatic solid tumors.
  Interventions: Drug: retifanlimab

INTERVENTIONS:
Drug: retifanlimab — Anti-PD-1 monoclonal antibody
  Other Names: INCMGA0012

SUMMARY:
The primary goal of this Phase 1 study is to characterize the safety and tolerability of INCMGA00012 and establish the maximum tolerated dose (MTD) of INCMGA00012 administered on either every two week or every four week schedules of administration among patients with solid tumors. Pharmacokinetics, pharmacodynamics, and the anti-tumor activity of INCMGA00012 will also be assessed.

The purpose of Amendment 5 is to obtain additional safety experience at the newly defined recommended Phase 2 dose of 500 mg every 4 weeks in patients with endometrial cancer, specifically either microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR). Additionally, every 3 week (Q3W) flat-dosing will be studied in an additional tumor agnostic cohort.

DETAILED DESCRIPTION:
This study is a Phase 1, open-label, dose escalation and cohort expansion study designed to characterize the safety, tolerability, PK, PD, immunogenicity, and preliminary anti-tumor activity of INCMGA00012 administered IV every 2, 3, or 4 weeks in patients with relapsed/refractory, unresectable locally advanced or metastatic solid tumors.

In the initial phase of the study, two dose schedules will be assessed in dose escalation, once every two weeks and once every four weeks administration of single agent INCMGA00012. Following the establishment of an MTD, additional patients will enroll in expansion cohorts of specific tumor types and/or INCMGA00012 dose.

The Cohort Expansion Phase will include tumor-specific cohorts, consisting of patients with endometrial cancer (unselected [up to n = 35] and MSI-H or dMMR [up to n = 70]), cervical cancer (up to n = 35), sarcoma (up to n = 35), non-small cell lung cancer (NSCLC) (up to n = 35), and 3 cohorts of any tumor histology (tumor-agnostic) (up to n = 15) who will receive flat dosing: 1 cohort treated with INCMGA00012 500 mg Q4W, 1 cohort with INCMGA00012 750 mg Q4W, and 1 cohort treated with INCMGA00012 375 mg Q3W.

ELIGIBILITY:
Inclusion Criteria:

Histologically proven, locally advanced unresectable or metastatic solid tumors for whom no approved therapy with demonstrated clinical benefit is available or standard treatment was declined. Patients enrolled to Cohort H (endometrial cancer 500 mg Q4W) must have MSI-H or dMMR endometrial cancer, as determined by a local laboratory using IHC or PCR methods and must also have tissue (fresh or archival) available for central confirmation of diagnosis

* Expansion cohort(s): Progression during or following at least 1, and up to 5, previous systemic therapies, consistent with the standard of care for the specific tumor type.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy ≥ 12 weeks
* Measurable disease
* Acceptable laboratory parameters

Exclusion Criteria:

* Symptomatic central nervous system (CNS) metastases.
* For Cohort Expansion, patients who have previously received an immune checkpoint inhibitor (e.g., anti-PD-L1, anti-PD-1, anti-CTLA-4) are not eligible for this study.
* Patients with any history of known or suspected autoimmune disease with the specific exceptions of vitiligo, resolved childhood atopic dermatitis, psoriasis not requiring systemic treatment (within the past 2 years), and patients with a history of Grave's disease that are now euthyroid clinically and by laboratory testing.
* Treatment with any systemic anti-neoplastic therapy, or investigational therapy within the 4 weeks prior to the initiation of study drug administration.
* Treatment with radiation therapy within 2 weeks prior to the initiation of study drug administration.
* Clinically significant cardiovascular disease
* Clinically significant pulmonary compromise, including a requirement for supplemental oxygen use to maintain adequate oxygenation.
* Presence of active pneumonitis or history of non-infectious pneumonitis.
* Clinically significant gastrointestinal disorders
* Evidence of active viral, bacterial, or systemic fungal infection requiring parenteral treatment within 7 days prior to the initiation of study drug. Patients requiring any systemic antiviral, antifungal, or antibacterial therapy for active infection must have completed treatment no less than one week prior to the initiation of study drug
* Known history of positive testing for human immunodeficiency virus or history of acquired immune deficiency syndrome.
* Known history of hepatitis B or hepatitis C infection or known positive test for hepatitis B surface antigen, hepatitis B core antigen, or hepatitis C polymerase chain reaction (PCR)
* Vaccination with any live virus vaccine within 4 weeks prior to the initiation of study drug administration. Inactivated annual influenza vaccination is allowed
* Dementia or altered mental status that would preclude understanding and rendering of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v4.03 | 24 months
  Safety is based on evaluation of adverse events (AEs) and serious adverse events (SAEs) from the time of study drug administration through the End of Study visit.
MTD | 24 months
  Maximum Tolerated Dose of INCMGA00012

SECONDARY OUTCOMES:
AUC | 24 months
  Area Under the Plasma Concentration versus Time Curve of INCMGA00012
Cmax | 24 months
  Maximum Plasma Concentration of INCMGA00012
Tmax | 24 months
  Time to reach maximum (peak) plasma concentration of INCMGA00012
Ctrough | 24 months
  Trough plasma concentration of INCMGA00012
Total body clearance of the drug from plasma (CL) of INCMGA00012 | 24 months
Vss | 24 months
  Apparent volume of distribution at steady state of INCMGA00012
t1/2 | 24 months
  Terminal half-life of INCMGA00012
ADA | 24 months
  Percent of patients with anti-drug antibody

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (80):
- United States (8):
  - Honor Health Research Institute, Scottsdale, Arizona
  - South Texas Accelerated Research Therapeutics, Grand Rapids, Michigan
  - Rutgers Cancer Institute of Nj, New Brunswick, New Jersey
  - Carolina Bio-Oncology Institute, Pllc, Huntersville, North Carolina
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Md Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
- Australia (2):
  - Chris Obrien Lifehouse, Camperdown, New South Wales
  - St Vincent'S Hospital Sydney, Darlinghurst, New South Wales
- Belgium (2):
  - Universitair Ziekenhuis (Uz) Leuven, Leuven
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
- Bulgaria (4):
  - COMPLEX ONCOLOGY CENTER ï¿½ BURGAS EOOD, Burgas
  - Mc Women'S Health-Nadezhda Eood, Sofia
  - Acibadem Cityclinica Mhat Tokuda, Sofia
  - Umhat in Oncology, Sofia
- China (17):
  - Peking Union Medical College Hospital, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Beijing Cancer Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Xiangya Hospital Central South University, Changsha
  - Hunan Cancer Hospital, Changsha
  - Sun Yat-Sen Memorial Hospital Sun Yat-Sen University, Guangzhou
  - The First Affiliated Hospital Sun Yat-Sen University, Guangzhou
  - Qilu Hospital of Shandong University, Jinan
  - Yunnan Cancer Hospital, Kunming
  - Zhongda Hospital Southeast University, Nanjing
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - The Second Hospital of Shanxi Medical University, Taiyuan
  - Tongji Hospital Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Henan Cancer Hostipal, Zhengzhou
- Finland (2):
  - Docrates Cancer Center, Helsinki
  - Turku University Hospital, Turku
- France (8):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - Centre Antoine Lacassagne, Nice
  - Hospital Universitaires de Geneve, Paris
  - Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris
  - Centre de Lutte Contre Le Cancer - Institut de Cancerologie de L'Ouest - Rene Gauducheau, Saint-Herblain
  - Universitaire Du Cancer de Toulouse Institut Claudius Regaud Iuct-Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (7):
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
  - CHARITE - UNIVERSITï¿½TSMEDIZIN BERLIN, Berlin
  - University Clinic Carl Gustav Carus Technical University Dresden, Dresden
  - Universitatsklinikum Essen, Essen
  - University Medical Center Freiburg, Freiburg im Breisgau
  - University Hospital Grosshadern Munich, Munich
  - STADTISCHE KLINIKUM MUNCHEN ï¿½ NEUPERLACH KLINIK FUR HAMATOLOGIE UND ONKOLOGIE, München
- Italy (4):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Ancona
  - Fondazione Del Piemonte Per L'Oncologia Ircc Candiolo, Candiolo
  - Istituto Nazionale Tumori Irccs Fondazione Pascale, Naples
  - Policlinico Universitario Agostino Gemelli Universita Cattolica Del Sacro Cuore, Rome
- Riga East University Hospsital, Riga, Latvia
- National Cancer Institute, Vilnius, Lithuania
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Wellington Hospital, Wellington
- Poland (9):
  - SZPITALE WOJEWï¿½DZKIE W GDYNI SPï¿½LKA Z OGRANICZONA ODPOWIEDZIALNOSCIA, Gdynia
  - University Hospital Krakow, Department of Oncology, Krakow
  - Ko-Med Centra Kliniczne Osrodek Badan Klinicznych W Lublinie, Lublin
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Msw Z W-McO W Olsztynie, Olsztyn
  - Biovirtus Research Site, Otwock
  - Szpital Kliniczny Przemienienia Panskiego, Poznan
  - Katedra I Klinika Onkologii Um W Poznaniu Oddzial Ginekologii Onkologicznej, Poznan
  - Medical University of Warsaw - 2Nd Department Obstetric and Gynecology, Warsaw
  - Centrum Onkologii - Instytut Im. Marii Sklodowskiej - Curie, Warsaw
- Spain (5):
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de La Paz, Madrid
  - Centro Integral Oncologico Clara Campal (Ciocc), Madrid
- Ukraine (5):
  - Multifield Clinical Hospital No 4, Dnipro
  - Regional Clinical Oncology Center Facility of State Higher Educational Institution, Ivano-Frankivsk
  - Rmi Sumy Regional Clinical Oncology Dispensary, Sumy
  - Uzhgorod National University Clinical Base Uzhgorod Central City Clinical Hospital, Uzhhorod
  - Podillia Regional Center of Oncology - Chemotherapy Department, Vinnytsia
- United Kingdom (3):
  - Sarah Cannon Research Institute, London
  - The Christie Nhs Foundation Trust Uk, Manchester
  - The Royal Marsden Nhs Foundation Trust - Chelsea, Sutton

IPD SHARING:
Plan to Share IPD: No